CLINICAL TRIAL: NCT04031079
Title: Use of Wearable Tech to Increase Physical Activity in Inpatient Rehabilitation for Overweight and Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/799
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Overweight
Keywords: Weight Loss; Rehabilitation; Exercise; Biomedical Technology
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: A parallel group design with two groups
Who Masked: Investigator
Masking Description: The researchers performing the analyses will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable tech with feedback (Experimental): This group will be wearing an activity measurement device (wristband) and receive feedback about their activity level through a mobile application while taking part in a traditional inpatient rehabilitation program for overweight and obesity (lifestyle change program).
  Interventions: Device: Wearable tech with feedback; Behavioral: Rehabilitation program
- Wearable tech without feedback (Active Comparator): This group will be wearing the same the activity measurement device as the intervention group, but they will not receive any feedback about their activity level. They will not have access to the mobile application. They will take part in the same rehabilitation program as the intervention group.
  Interventions: Device: Wearable tech without feedback; Behavioral: Rehabilitation program

INTERVENTIONS:
Device: Wearable tech with feedback — an armwrist device measuring physical activity level. The user will receive information about their physical activity level through their smartphone
  Arms: Wearable tech with feedback
Device: Wearable tech without feedback — an armwrist device measuring physical activity level, no reporting back to the user
  Arms: Wearable tech without feedback
Behavioral: Rehabilitation program — traditional inpatient rehabilitation program for overweight and obesity (lifestyle change program)

SUMMARY:
The aim of this project is to evaluate whether use of wearable tech increases physical activity in patients participating in inpatient rehabilitation for overweight and obesity.

DETAILED DESCRIPTION:
Obesity is a global epidemic with profound consequences for individuals and societies. Physical exercise is important for weight reduction and weight loss maintenance. Use of wearable tech might facilitate physical activity. Here it will be evaluated whether use of wearable tech that gives feedback about the user's activity level, increases physical activity in people participating in inpatient rehabilitation for overweight and obesity. The control group will be wearing the same wearable tech as the intervention group, but they will not receive any feedback about their activity level.

The feedback application will give participants in the intervention group information about the number of PAI they earn each week. PAI is short for Personal Activity Intelligence. One earns PAI points every time heart rate increases: The higher heart rate, the faster one earns PAI. Previous research have shown that those who achieve 100 PAI or more every week over time, live for an average of more than eight years longer than others.

During the study all participants will take part in a traditional inpatient rehabilitation program (lifestyle modification program). The program consist of three periods at the rehabilitation center with time at home in-between. The study will take place during two periods at the center and one period at home. Time spent on physical activity and number of earned PAI's will be counted during the period at home.

ELIGIBILITY:
Inclusion Criteria:

* taking part in inpatient rehabilitation at Unicare Helefort Rehabilitation center for overweight or obesity.
* having been referred from a hospital outpatient obesity clinic.

Exclusion Criteria:

* not having a smartphone (will not be able to access the mobile application).
* using a wheelchair (the technology will be not able to measure activity correctly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Activity level | 4 weeks (time period at home between two stays at the rehabilitation center)
  Time spent in moderate to vigorous physical activity (minutes per day)
Number of PAIs | 4 weeks (time period at home between two stays at the rehabilitation center)
  mean number of Personal Activity Intelligence (PAI) points achieved per week
Percentage achieving 100 Personal Activity Intelligence points (PAIs) per week | 4 weeks (time period at home between two stays at the rehabilitation center)

SECONDARY OUTCOMES:
oxygen uptake | 7 weeks (from inclusion to end of rehabilitation program)
  submaximal oxygen uptake measured by the Astrand bicycle test (described in Textbook of work physiology by Astrand from 1986)
Body weight | 7 weeks (from inclusion to end of rehabilitation program)
  body weight in kilograms
Body Mass Index score | 7 weeks (from inclusion to end of rehabilitation program)
  weight in kilograms divided by height in metres squared

CONTACTS AND LOCATIONS:
Overall Officials: Lene Aasdahl, PhD MD, Principal Investigator — National Taiwan Normal University; Jorunn Helbostad, Dr Philos, Study Director — Norwegian University of Science and Technology
Locations (1):
- Unicare Helsefort, Rissa, Norway

IPD SHARING:
Plan to Share IPD: No